CLINICAL TRIAL: NCT05818345
Title: Socioeconomic Position and the Effectiveness of a Pricing Intervention Based on Energy Content in Restaurants: a Real-world Experiment
Brief Title: Pricing Interventions Based on Energy Content in Restaurants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Restaurant has closed down
Sponsor: University of Liverpool (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Eric Robinson, Professor, University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Restaurant Study
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Healthy Diet; Eating Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive a standard menu with the existing pricing structure of the restaurant
- Pricing Intervention (Experimental): Participants will receive a menu where lower kcal dishes are discounted by 30%
  Interventions: Behavioral: Pricing intervention

INTERVENTIONS:
Behavioral: Pricing intervention — Participants will be provided with a menu with manipulated prices for products with lower kilocalories
  Arms: Pricing Intervention

SUMMARY:
The goal of this clinical trial is to examine the impact of price decreases based on energy content in a full-service restaurant on immediate dietary consumption (in terms of kilocalories (kcals), sugar, fat, and salt intake) and dietary consumption the rest of the day following the intervention; and whether the intervention effects differ based on socioeconomic position (SEP).

Participants will be asked to visit the restaurant twice. At visit 1, participants will receive a control study menu with the existing pricing structure of the restaurant. At visit 2, participants will receive the same study menu with the pricing intervention introduced.

For comparative purposes a smaller subgroup of participants will receive the control menu at both visit 1 and 2 to allow the researchers to estimate whether any pre-post changes occur in the absence of a pricing intervention (and whether change differs by SEP).

ELIGIBILITY:
Inclusion Criteria:

* UK resident, aged 18 and older, fluent in English, have an out-of-home meal at least once a month and have no dietary allergies

Exclusion Criteria:

* No further exclusion criteria as it is a real-world study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Total kilocalories (kcal) ordered at the restaurant | 1 hour
  The researchers will observe whether the total kcal ordered is different with a standard menu versus the menu with price manipulations
Total kcal consumed at the restaurant | 1 hour
  The researchers will observe whether the total kcal consumed (taking into account leftovers and food sharing) is different with a standard menu versus the menu with price manipulations

SECONDARY OUTCOMES:
Later kcal intake | 10 hours
  The researchers will examine dietary intake the rest of the day following the restaurant visit to examine evidence of compensatory dietary intake.
Total sugar, fat and salt intake | 1 hour
  The researchers will observe whether the total sugar, fat and salt ordered is different with a standard menu versus the menu with price manipulations

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Liverpool, Liverpool, Merseyside
  - University of Liverpool, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On publication, indefinitely